CLINICAL TRIAL: NCT03204240
Title: Targeting Skeletal Muscle to Improve Metabolic Health in Individuals With Spinal Cord Injury (SCI)
Brief Title: Metabolic Health in Individuals With Spinal Cord Injury (SCI)
Acronym: SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Ceren Yarar-Fisher, Principal Investigator, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 000512788
Record Dates: First submitted 2017-06-14; First posted 2017-06-29 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Spinal Cord Injuries; Skeletal Muscle Atrophy; Metabolic Disease
Keywords: Spinal Cord Injury; Skeletal Muscle; Functional Electrical Stimulation; Diabetes
MeSH Terms: conditions — Spinal Cord Injuries; Muscular Atrophy; Metabolic Diseases; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This group will receive electrical stimulation induced exercises in addition to their standard care during in-patient rehabilitation (IPR). Standard care will include respiration therapy, bed mobility, transfers, wheelchair mobility skills, bowel and bladder management, tone and spasticity management, and skills for performing other activities of daily living. Exercises will include neuromuscular electrical stimulation (NMES) induced-resistance exercise (RE) (1x/day) and NMES-aerobic exercise (1x/day) for 3 days/week.
  Interventions: Other: Neuromuscular electrical stimulation
- Control (No Intervention): This group will receive standard care plus passive dynamic exercise of the lower legs (sham treatment for NMES-RE, 1x/day) and transcutaneous electrical nerve stimulation (TENS, sham treatment for NMES-aerobic exercise, 1x/day) during IPR.

INTERVENTIONS:
Other: Neuromuscular electrical stimulation — NMES-RE will involve concentric/eccentric contractions of the quadriceps from a seated position. Briefly, each session will include four sets of 10 actions evoked using 50 Hz trains of 450 µs biphasic pulses. The protocol will be implemented using surface NMES. Upon completion of the NMES-RE session, participants will be given a short break (10-15 minutes) for recovery before starting aerobic training. NMES aerobic exercise will involve twitch electrical stimulation (pulse duration/interval=200/50 µs) applied to the quadriceps muscle via surface NMES. The current amplitude will set to 175 mA. The training will start with 10 minutes of twitch stimulation at 2 Hz. After the first weeks, the duration of the session will progressively increase up to 60 minutes at 10 Hz.
  Arms: Intervention

SUMMARY:
Individuals with spinal cord injury (SCI) live longer than before and live to an age where metabolic disorders become highly prevalent. Due to loss of mobility and severe skeletal muscle atrophy, obesity, glucose intolerance, and peripheral insulin resistance develop soon after the onset of SCI. These abnormalities are thought to contribute to the increased diabetes disease risk and accelerated aging process in the SCI population. As a result of these trends, overall burden of complications, economic impact and reduced quality of life are increasing. Until there are effective treatments for SCI, it is imperative to develop effective interventions to mitigate metabolic disorders that develop in individuals with SCI. The proposed research project examines the impact of early utilization of a novel neuromuscular electrical stimulation (NMES) program on skeletal muscle metabolism and overall metabolic health in individuals with sub-acute, complete SCI.

DETAILED DESCRIPTION:
The escalating prevalence of metabolic disorders in individuals with long-standing spinal cord injury (SCI) highlights the urgent need for early interventions for prevention and improving quality of life. Individuals with SCI, while often relatively young, are at high risk for developing insulin resistance and type 2 diabetes soon after the onset of injury. Skeletal muscle is the major site of dietary glucose disposal, yet the relationship between adaptations in skeletal muscle after SCI and the development of metabolic disturbances remains poorly understood. Within 6 months after SCI, lower limb muscles atrophy by up to 45% and individuals show a 3-fold increase in intramuscular fat levels compared to able-bodied (AB) controls. Moreover, within 6 months after SCI, fatigue-resistant and oxidative Type I and Type IIa muscle fibers transform into highly fatigable, glycolytic Type IIax and IIx muscle fibers with impaired oxidative metabolism. The maintenance of adequate muscle mass and metabolic function has never been targeted as a potential strategy to prevent chronic metabolic disorders in individuals with SCI. Early prevention of these deleterious adaptations is expected to be more effective than attempting to reverse changes several months or years after SCI.

Among the available experimental strategies to reverse atrophy and improve skeletal muscle metabolism in individuals with SCI, there seems to be consensus that muscle contraction via neuromuscular electrical stimulation (NMES) is the most potent approach. The investigators recently showed that 8 weeks of NMES-resistance exercise in people with long-standing SCI effectively increased myofiber size and distribution of Type IIa myofibers; however, this intervention did not increase the distribution of Type I fibers. There is a need for novel NMES programs that induce key molecular adaptations to both resistance and aerobic exercise to maintain an oxidative, fatigue-resistant, and insulin-sensitive phenotype following SCI.

Here, the investigators propose an early intervention of combined NMES (Comb-NMES). This program couples electrically induced resistance and aerobic exercise on the knee extensor muscle group (quadriceps) with the goal of maintaining or even improving muscle mass and metabolic function. The proposed Comb-NMES program repetitively stresses the paralyzed knee extensor muscles with both low frequency electrical stimulation (aerobic training) to improve oxidative metabolism and retain Type I fibers and high frequency (resistance training) electrical stimulation with dynamic contractions to prevent atrophy and retain Type IIa fibers.

The investigators will test the following central hypothesis that, compared to a control group, those treated with Comb-NMES for 6 weeks early after SCI will maintain a better whole-body metabolic profile, largely driven by maintenance of paralyzed muscle mass, fiber phenotype (maintenance of Type I and IIa fibers), and muscle oxidative metabolic function. The investigators will test this hypothesis in a controlled clinical trial of patients with SCI with the following specific aims:

Aim 1: Quantify the effects of Comb-NMES on clinically important measures of metabolic function.

Hypothesis 1. Compared to a control group, 6 weeks of Comb-NMES (3 days/week) will maintain higher glucose tolerance and whole-body insulin sensitivity.

Aim 2: Quantify cellular, molecular and functional adaptations in the quadriceps muscle that are responsible for improvements in muscle metabolism and overall metabolic profile.

Hypothesis 2.1. Compared to a control group, 6 weeks of Comb-NMES (3 days/week) will maintain better muscle glucose utilization, oxidative metabolism, muscle size, strength, and fatigue resistance, as well as a healthy muscle fiber phenotype (homogeneous distribution of Type I, IIa, and IIx fibers).

Hypothesis 2.2. Comb-NMES-induced improvements in overall metabolic profile will be reflected in changes in metabolite signatures related to muscle mitochondrial function and intermediary metabolism.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 and 60 years;
* diagnosis of traumatic SCI at the cervical or thoracic level (C5-T12) classified as AIS A (motor and sensory complete);
* within 14 days of the SCI and the first week of initial inpatient rehabilitation;
* medically stable at the time of testing;
* no history of metabolic syndrome and/or type 1 or type 2 diabetes.

Exclusion Criteria:

* Pregnant women
* Orthopedic condition that limits lower extremity function
* Neurological (other than SCI), vascular, or cardiac problems that may limit function and interfere with testing procedures
* Have 1 or more contraindications to NMES
* Have lidocaine or iodine allergy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity | Week1 and Week 6 of IPR
  Liquid meal test will be given and blood samples will be collected before and after meal ingestion.
Change in glucose tolerance | Week 1 and Week 6 of IPR
  Liquid meal test will be given and blood samples will be collected before and after meal ingestion.
Change in beta cell function | Week 1 and Week 6 of IPR
  Liquid meal test will be given and blood samples will be collected before and after meal ingestion.

SECONDARY OUTCOMES:
Change in metabolic signaling in skeletal muscle | Week1 and Week 6 of IPR
  Muscle samples will be collected via our established percutaneous needle biopsy procedure.
Change in muscle strength | Week 1 and Week 6 of IPR
  The quadriceps femoris muscle group will be studied during NMES-elicited muscle contractions both in the intervention and control groups.
Change in muscle fatigue | Week 1 and Wekk 6 of IPR
  The quadriceps femoris muscle group will be studied during NMES-elicited muscle contractions both in the intervention and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ceren Yarar-Fisher, PhD, Principal Investigator — OSU
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided